CLINICAL TRIAL: NCT01935648
Title: Blood Levels of Local Anaesthetic in Knee Arthroplasty: A Pharmacological Study of Ropivacaine Blood Levels During the Caledonian Technique for Knee Arthroplasty
Brief Title: Blood Levels of Local Anaesthetic in Knee Arthroplasty Using a Continuous Infusion Device
Acronym: BLOCKS-II
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: B. Braun Medical Inc. (Industry); University of Strathclyde (Other)
Responsible Party: Sponsor
Other Study IDs: 13/ANAES/02
Record Dates: First submitted 2013-07-29; First posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Up to 11 blood samples per patient
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ropivacaine: Injection of local anaesthetic (ropivacaine) into the knee joint following hip arthroplasty. Total dose 200mls of 0.2% ropivacaine or 400mg at the time of surgery. This will be followed by a continuous infusion of 10mls/hour 0.2% ropivacaine for the subsequent 24 hours.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine
  Other Names: Naropin

SUMMARY:
The primary goal is to evaluate ropivacaine blood concentrations during and after local anaesthetic (ropivacaine) infiltration - the Caledonian technique - for total knee replacement surgery. The investigators plan to measure these levels by testing blood samples taken over a timed period.

This will allow us to confirm whether the current regimen of local anaesthetic use is within safe limits.

DETAILED DESCRIPTION:
Local anaesthetic (LA) toxicity may occur when the blood levels of a drug become particularly high. There is a need to confirm that the technique is safe to use. In addition, journal case reports may only describe serious side-effects of toxicity such as abnormal heart rhythms whilst more subtle clinical signs are rarely reported.

The investigators would like to study whether or not toxic levels may be approached in some patients or whether more subtle toxicity symptoms and signs are missed. For example, irregular heartbeat, low blood pressure or confusion/agitation.

Therefore, the investigators intend to study ropivacaine blood levels in patients receiving a total hip replacement in the Golden Jubilee National Hospital. A series of timed samples will be taken during the perioperative period. The anaesthesia and surgery will be performed as routine and no new treatment will be involved. Patient demographics, ropivacaine blood levels and clinical observations following LA administration will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients greater than 65 years of age

Exclusion Criteria:

* Patients with a known sensitivity/allergy to ropivacaine or amide-type local anaesthetics
* Patients who are not suitable for the Caledonian technique
* Patients who refuse or are unable to give consent
* Patients undergoing bilateral hip replacements
* Patients with known heart, liver or kidney failure

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients undergoing elective knee joint replacement where they will be receiving the Caledonian technique
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of ropivacaine | Start of surgery until 24 hours postoperatively
  Plasma levels of ropivacaine will be analysed to determine total and free levels. These will be taken following tourniquet release at the following time points:
  5, 10, 15, 20, 25, 30 minutes then 1, 4, 12 and 24 hours. Note: Each patient will also have a baseline blood sample taken.

SECONDARY OUTCOMES:
Vital signs of heart rate and blood pressure | Start of surgery until 24 hours postoperatively
  Vital signs will be recorded (at each time point) when blood samples are taken.
Continuous 24 hour electrocardiograph monitoring | First 24 hours after surgery
  Electrocardiograph data will be reported using analysis software to provide a summary of heart rhythm over the study period. Both minor abnormalities (ectopic beats) and major abnormalities (loss of sinus rhythm, heart block) will be detected and reported.
Symptoms of local anaesthetic toxicity | Start of surgery until 24 hours postoperatively
  Patients will be specifically questioned (at each time point) on whether they have any of the following symptoms:
  Perioral tingling, dizziness, blurred vision, nausea
Signs of local anaesthetic toxicity | Start of surgery until 24 hours postoperatively
  Patients will be specifically assessed (at each time point) for the following signs:
  Confusion/agitation, (loss of consciousness, seizure activity, cardiac arrest)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gill, MBChB, Principal Investigator — NHS Research Scotland
Locations (1):
- Golden Jubilee National Hospital, Clydebank, West Dunbartonshire, United Kingdom